CLINICAL TRIAL: NCT03213964
Title: Intraperitoneal Delivery of Adaptive Natural Killer (NK) Cells (FATE-NK100) With Intraperitoneal Interleukin-2 in Women With Recurrent Ovarian, Fallopian Tube, and Primary Peritoneal Cancer
Brief Title: Intraperitoneal Delivery of Adaptive Natural Killer (NK) Cells (FATE-NK100) With Intraperitoneal Int
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016LS186
Record Dates: First submitted 2017-07-07; First posted 2017-07-11 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Epithelial Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Cancer
Keywords: Recurrent; Platinum Resistant; Platinum Sensitive
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms; Recurrence | interventions — Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): FATE-NK100 is a donor-derived NK cell product comprising ex vivo activated effector cells with enhanced anti-tumor activity.
  FATE-NK100 is administered to determine the maximum tolerated doze/maximum feasible dose (MTD/MFD).
  Interleukin-2 (IL-2) remains the only FDA approved drug that is capable of promoting NK cells activation and survival.
  Lymphodepletion with Cyclophosphamide and Fludarabine.
  Interventions: Biological: FATE-NK100; Drug: Interleukin-2

INTERVENTIONS:
Biological: FATE-NK100 — FATE-NK100 Infusion (Day 0)
  The FATE-NK100 product will be placed in approximately 100 cc of 5% human serum albumin.
  * Dose Level 1: 1 x 10^7 cells/kg IP
  * Dose Level 2: >1x10^7 cells/kg to ≤3x10^7 cells/kg
  * Dose Level 3: Complete FATE-NK100 bag (≥3 x 10^7 to ≤ 10 x 10^7 cells/kg)
Drug: Interleukin-2 — Interleukin-2 (begin Day 0): 6 million units three times a week for a total of 6 doses. For patients weighing less than 45 kilograms, the IL-2 will be given at 3 million units/m2 three times a week for 6 doses.
  The 1st dose will be given immediately (within 30 minutes) after the FATE-NK100 cell infusion on Day 0 as an inpatient. The remaining doses will be given in an outpatient setting.
  Other Names: IL-2

SUMMARY:
This is a Phase I trial to determine the maximum tolerated dose/maximum feasible dose (MTD/MFD) of a single infusion of FATE-NK100 via intra-peritoneal catheter in women with recurrent ovarian, fallopian tube or primary peritoneal cancer meeting one of the following minimal prior treatment requirement:

* Platinum resistant: may receive FATE-NK100 as 2nd line (as 1st salvage therapy). Platinum resistant is defined as disease that has responded to initial chemotherapy but demonstrates recurrence within a relatively short period of time (< 6 months) following the completion of treatment.
* Platinum sensitive: may receive FATE-NK100 as 3rd line therapy (as 2nd salvage therapy). Platinum sensitive is defined as the recurrence of active disease in a patient who has achieved a documented response to initial platinum-based treatment and has been off therapy for an extended period of time (≥ 6 months).

ELIGIBILITY:
Inclusion Criteria:

* Recurrent epithelial ovarian cancer, fallopian tube, or primary peritoneal cancer meeting one of the following minimal prior treatment requirement (no limit to the maximum number of prior treatments):

  * Platinum Resistant: may receive FATE-NK100 as 2nd line (as 1st salvage therapy) with platinum resistant is defined as disease that has responded to initial chemotherapy but demonstrates recurrence within a relatively short period of time (< 6 months) following the completion of treatment.
  * Platinum Sensitive: may receive FATE-NK100 as 3rd line therapy (as 2nd salvage therapy) with platinum sensitive is defined as the recurrence of active disease in a patient who has achieved a documented response to initial platinum-based treatment and has been off therapy for an extended period of time (≥ 6 months).
* Measurable disease per RECIST within the abdomen and pelvis. Extra-peritoneal disease is permitted; however each lesion must be < 5 cm at the largest diameter.
* Available HLA haploidentical or better but not fully HLA-matched (2/4 or 3/4 antigens) related donor (aged 18 to 75 years) with donor/recipient match based on a minimum of intermediate resolution DNA based Class I typing of the A and B locus who is CMV seropositive.
* At least 18 years of age, but not older than 75 years
* GOG Performance Status 0, 1, or 2
* Adequate organ function within 14 days of study registration (28 days for pulmonary and cardiac) defined as:

  * Hematologic: platelets ≥ 80,000 x 109/L and hemoglobin ≥ 9 g/dL, unsupported by transfusions; absolute neutrophil count (ANC) ≥ 1000 x 109/L, unsupported by G-CSF or granulocytes
  * Creatinine: Estimated glomerular filtration rate (eGFR) ≥ 50 mL/min/1.73m2 per current institutional calculation formula
  * Hepatic: AST and ALT ≤ 3 x upper limit of institutional normal
  * Pulmonary Function: Oxygen saturation ≥ 90% on room air; PFT's required only if symptomatic or prior known impairment - must have pulmonary function >50% corrected DLCO and FEV1
  * Cardiac Function: LVEF ≥ 40% by echocardiography, MUGA, or cardiac MRI; no uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities

Exclusion Criteria:

* Able to be off prednisone or other immunosuppressive medications for at least 3 days prior to FATE-NK100 cell infusion (excluding preparative regimen pre-medications)
* Agrees to the placement of an intraperitoneal port before the start of chemotherapy and remains in place through Day 28 or longer
* Washout period of at least 14 days after any approved or experimental tumor directed therapy prior to start of cyclophosphamide and fludarabine
* If history of brain metastases must be stable for at least 3 months after treatment - A brain CT scan or MRI is only be required in subjects with known brain metastases at the time of enrollment or in subjects with clinical signs or symptoms suggestive of brain metastases
* Voluntary written consent prior to the performance of any research related procedures

Exclusion Criteria:

* Untreated brain metastases
* Myocardial Infarction (MI) within the previous 6 months
* Active autoimmune disease requiring systemic immunosuppressive therapy
* History of severe asthma and currently on chronic systemic medications (mild asthma requiring inhaled steroids only is eligible)
* New or progressive pulmonary infiltrates on screening chest X-ray or chest CT scan unless cleared for study by Pulmonary. Infiltrates attributed to infection must be stable/improving (with associated clinical improvement) after 1 week of appropriate therapy (4 weeks for presumed or documented fungal infections).
* Uncontrolled bacterial, fungal or viral infections with progression of clinical symptoms despite therapy
* Known history of HIV positivity or active hepatitis C or B - chronic asymptomatic viral hepatitis is allowed
* Received any investigational agent within the 14 days before the start of study treatment (1st dose of fludarabine)
* Disease outside of the peritoneal cavity

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-10-19 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-03-10 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Doze of FATE-NK100 | 1 Year
  To determine the maximum tolerated dose/maximum feasible dose (MTD/MFD) of FATE-NK100 when administered via intraperitoneal catheter in patients with recurrent ovarian, fallopian tube, and primary peritoneal cancer.

SECONDARY OUTCOMES:
Objective Response Rate | Day 28
  Incidence of objective response rate (ORR) of the FATE-NK100 treatment
Progression-Free Survival (PFS) | 6 Months
  Incidence of progression-free survival of treated patients 6 months post-infusion
Overall Survival (OS) | 6 Months
  Incidence of overall survival of treated patients 6 months post-infusion

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Geller, MD, MS, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States